CLINICAL TRIAL: NCT04650659
Title: Measurement Properties and Performance of Functional Exercise Tests in Patients With Systemic Sclerosis
Brief Title: Functional Exercise Tests in Patients With Systemic Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Rheumatism Association (Other)
Responsible Party: Sponsor
Other Study IDs: SSc6MWT2020; 1-16-02-270-20 (Other: The Danish Data Protection Agency)
Record Dates: First submitted 2020-11-23; First posted 2020-12-03 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Scleroderma, Systemic; Lung Diseases, Interstitial; Pulmonary Arterial Hypertension; Acroosteolysis
Keywords: 6-Minute Walk Test; Scleroderma, Systemic; Oximetry; Exercise test; Raynaud Disease; HR-pQCT; Nailfold videocapillaroscopy
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial; Pulmonary Arterial Hypertension; Acro-Osteolysis; Raynaud Disease | interventions — Microscopic Angioscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1 mL arterial blood will be drawn from an arterial line before and after the 6MWT, respectively. In total 2 mL of arterial blood. Blood gas analysis will be performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Part one of the project: 83 patients with Systemic Sclerosis will perform three functional exercise tests on the same day. All 83 patients will be examined with NVC. Moreover, HRpQCT will be performed on all patients at baseline and after 1 year.
  Interventions: Diagnostic Test: 6-minute walk test part one; Diagnostic Test: 1-minute sit-to-stand test; Diagnostic Test: 4-meters gait speed test; Diagnostic Test: Nailfold videocapillaroscopy; Diagnostic Test: HR-pQCT; Diagnostic Test: Hand x-ray; Diagnostic Test: DEXA
- Part two of the project: Half of the patients from part one of the project will be invited to repeat the three functional exercise tests approximately one week later in reverse order to determine test-retest reliability.
  Interventions: Diagnostic Test: 6-minute walk test part two; Diagnostic Test: 1-minute sit-to-stand test; Diagnostic Test: 4-meters gait speed test

INTERVENTIONS:
Diagnostic Test: 6-minute walk test part one — Measurement of: 6-minute walk distance, the modified Borg scale before and after testing and continuous measure of peripheral oxygen saturation and heart rate. The peripheral oxygen saturation will be measured continuously on three anatomical location: the forehead, an earlobe and a finger. In patients who will accept an arterial line will be placed and blood gas will be analyzed.
  Groups: Part one of the project
Diagnostic Test: 6-minute walk test part two — Measurement of: 6-minute walk distance, the modified Borg scale before and after testing and continuous measure of peripheral oxygen saturation and heart rate. The peripheral oxygen saturation will be measured continuously on three anatomical location: the forehead, an earlobe and a finger. No arterial line will be placed.
  Groups: Part two of the project
Diagnostic Test: 1-minute sit-to-stand test — Measurement of: Number of repetitions, the modified Borg scale before and after testing and continuous measure of peripheral oxygen saturation and heart rate. The peripheral oxygen saturation will be measured on the three anatomical locations mentioned above.
Diagnostic Test: 4-meters gait speed test — Measurement of: Time to complete the 4 meters course and calculation of the 4-meters-gait-speed.
Diagnostic Test: Nailfold videocapillaroscopy — Capillary density measurement of: The finger with the probe and the average of all the fingers.
  NVC with 200 x magnification will be performed on the 2nd to 5th finger on both hands.
  Groups: Part one of the project
Diagnostic Test: HR-pQCT — Imaging: One arm is scanned in a 9 mm-long volume of the distal radius (110 slices), and the distal part of the 2nd to 5th finger on both hands are scanned in a 36,08 mm-long volume (440 slices) at baseline and after 1 year.
  Groups: Part one of the project
Diagnostic Test: Hand x-ray — Imaging: Hand x-ray was performed on patients scanned with HR-pQCT, unless images were already available (≤ 1 year).
  Groups: Part one of the project
Diagnostic Test: DEXA — Imaging: A bone density (DEXA) scan was performed on patients scanned with HR-pQCT, unless it was already available (≤ 2 years).
  Groups: Part one of the project

SUMMARY:
The aim of the study is to examine the validity of peripheral oxygen saturation measurement during the 6-minute walk test in patients with Systemic Sclerosis (SSc) and to examine the utility of two other functional tests as markers of pulmonary involvement in patients with SSc.

DETAILED DESCRIPTION:
Systemic Sclerosis (SSc) is a connective tissue disease characterized by progressive organ fibrosis and vascular dysfunction. The leading causes of disease related morbidity and mortality are interstitial lung disease (ILD) and pulmonary arterial hypertension (PAH). The 6-minute walk test (6MWT) is a submaximal functional exercise test used to evaluate ILD and PAH in patients with SSc. Desaturations during the 6MWT have been considered suggestive of ILD and PAH. Still, the optimal method to measure peripheral oxygen saturation during the 6MWT in patients with SSc remains unclear. Furthermore, other functional exercise tests may also be useful in patients with SSc.

Patients with SSc will perform three functional exercise tests, and approximately half of the patients will be invited to repeat the tests 1 week later to determine test-retest reliability. Additionally, nailfold videocapillaroscopy (NVC) will be performed on every patient to assess the capillary density of the nailfold of the fingers. Furthermore, to study the effect of SSc on bone, a high resolution peripheral quantitative computed tomography (HRpQCT) scan of radius and distal interphalangeal joints (DIP)/distal phalanges will be performed.

During the 6MWT, the peripheral oxygen saturation (SpO2) will be measured continuously on three anatomical locations. An arterial line will be placed, and blood will be drawn at baseline and after ended 6MWT and analysed for arterial oxygen saturation (SaO2). The correlation between the capillary density of the nailfold and the SpO2 measured on the finger will be assessed. The correlation between capillary density of the nailfold and bone status in the fingers and distal radius assessed with HRpQCT will be evaluated, and HRpQCT images will be compared with conventional radiography and DEXA. Bland-Altman plot will be used to display the agreement between SaO2 and SpO2 and between the two 6MWT. Further, the association between pulmonary variables and 6MWT results will be examined.

Two alternative functional exercise tests will be investigated and compared to results in the 6MWT: The 1-minute sit-to-stand test (1STST) and the 4-meter gait speed test (4MGS). The association between the three functional exercise tests and clinical parameters in patients with SSc will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Systemic Sclerosis according to the ACR/EULAR 2013 criteria
* Provided written informed consent

Exclusion Criteria:

* Overlap syndrome (except for rheumatoid arthritis and Sjögren syndrome)
* Recent or ongoing lung infection
* Other major comorbidities that could affect the functional exercise tests.
* Pregnancy
* Unable to understand the patient information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited if they have a clinical course at the Department of Rheumatology, Aarhus University Hospital (>500 patients with Scleroderma)
Sampling Method: Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Examine the validity of peripheral oxygen saturation measurement during 6-minute walk test in patients with Systemic Sclerosis. | 1 hour
  The agreement between the peripheral oxygen saturation measured on the forehead, finger and earlobe and the arterial oxygen saturation from the blood gas analysis will be examined.

SECONDARY OUTCOMES:
Examine the correlation between the 6-minute walk test, the 1-minute sit-to-stand test, and the 4-meter gait speed test in patients with Systemic Sclerosis. | 1 hour
  The agreement between the 6-minute walk test, the 1-minute sit-to-stand test, and the 4-meter gait speed test in patients with Systemic Sclerosis.
Investigate the correlation between functional exercise tests and the severity of pulmonary involvement in patients with Systemic Sclerosis. | 1 hour
  The agreement between functional exercise tests and the severity of pulmonary involvement in patients with Systemic Sclerosis.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Søndergaard, MD, PhD, Study Chair — Department of Rheumatology, Aarhus University Hospital, DK; Amanda Lynggaard Riis, Student, Principal Investigator — Department of Rheumatology, Aarhus University Hospital, DK; Esben Uggerby Næser, MD, PhD, Study Director — Department of Rheumatology, Aarhus University Hospital, DK; Katja Thorup Aaen, Student, Principal Investigator — Department of Rheumatology, Aarhus University Hospital, DK; Ellen-Margrethe Hauge, Professor, Study Chair — Department of Rheumatology, Aarhus University Hospital, DK; Frederik Cosedis Enevoldsen, Student, Principal Investigator — Department of Rheumatology, Aarhus University Hospital, DK; Rasmus Klose Jensen, MD, PhD, Study Director — Department of Rheumatology, Aarhus University Hospital, DK; Josephine Therkildsen, MD, Study Director — Department of Rheumatology, Aarhus University Hospital, DK
Locations (1):
- The Department of Rheumatology, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Elkjaer AL, Naeser EU, Aaen KT, Hovgaard HL, Juhl-Olsen P, Bendstrup E, Sondergaard K. Validity and reliability of measurement of peripheral oxygen saturation during the 6-Minute Walk Test in patients with systemic sclerosis. Rheumatol Int. 2024 Apr;44(4):611-620. doi: 10.1007/s00296-024-05532-5. Epub 2024 Feb 10. PMID 38340159